CLINICAL TRIAL: NCT02521831
Title: Neuroinflammatory and Neurocognitive Effects of Spinal vs. Inhalational Anesthesia for Elective Surgery in Infants: A Randomized, Controlled, Double-Blinded Study
Brief Title: Neuroinflammatory and Neurocognitive Effects of Spinal vs. Inhalational Anesthesia for Elective Surgery in Infants
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Emmett Whitaker, M.D. (Other)
Responsible Party: Sponsor-Investigator, Emmett Whitaker, M.D., Clinical Assistant Professor, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB15-00125
Record Dates: First submitted 2015-07-30; First posted 2015-08-13 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Inguinal Hernia
Keywords: Circumcision
MeSH Terms: conditions — Hernia, Inguinal | interventions — Anesthesia, Spinal; Bupivacaine; Anesthesia, Conduction; Anesthesia, General; Isoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- General Anesthesia (Active Comparator): Inhalational anesthesia with Isoflurane 1-2% in 50%/50% oxygen/air mixture.
  This arm will receive the General Anesthesia (isoflurane) intervention exclusively.
  Interventions: Drug: General Anesthesia (isoflurane)
- Spinal Anesthesia (Active Comparator): These infants will not receive any anesthetic gas prior to the spinal. These infants will be conscious for this procedure.
  Spinal will be administered, containing 0.25% isobaric bupivacaine, 1 mg/kg (maximum 5mg), Clonidine, 1 µg/kg, and Epinephrine, 1:200,000.
  This arm will receive the Spinal Anesthesia (bupivacaine) intervention exclusively.
  Interventions: Drug: Spinal Anesthesia (bupivacaine)

INTERVENTIONS:
Drug: Spinal Anesthesia (bupivacaine) — Bupivacaine is an amide-type, long-acting local anesthetic. Brand names include Exparel, Marcaine, and Sensorcaine.
  Other Names: Regional Anesthesia
  Arms: Spinal Anesthesia
Drug: General Anesthesia (isoflurane) — Isoflurane is a fluorinated ether with general anesthetic and muscle relaxant effects. Brand names include Forane and Terrell.
  Other Names: Standard Inhalational Anesthesia
  Arms: General Anesthesia

SUMMARY:
Significant concern regarding the safety of general anesthesia in children has arisen due to myriad animal studies suggesting neurotoxicity of commonly used anesthetic agents. Inflammation of the central nervous system after anesthesia may have a significant role in the pathogenesis of anesthetic-induced neural injury. To evaluate this hypothesis, the investigators propose to randomize healthy infants undergoing elective surgery to one of two anesthetics: 1) spinal anesthesia only; or 2) general inhalational anesthesia with isoflurane, laryngeal mask airway (LMA) or endotracheal tube (ETT), and single-shot caudal block. Primary endpoint will be serum inflammatory biomarkers and transcriptome analysis and secondary endpoint will be neurocognitive outcome at 6 months and 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Otherwise healthy child aged 0-less than 13 months undergoing elective (non-emergent) general, urologic, orthopedic, and plastic surgery
2. Parent/guardian must provide written informed consent in accordance with human investigation committee guidelines
3. Participants must be American Society of Anesthesiologist (ASA) physical status ≤ 2

Exclusion Criteria:

1. Any active bacterial or viral infection within the last 14 days
2. Treatment in the last 48 hours with non-steroidal anti-inflammatory (NSAID) or corticosteroid medications, or any other drug known to suppress or induce inflammation
3. Anticoagulant administration in the last 48 hours
4. Patients that have an American Society of Anesthesiologists physical status >2
5. Infants born more than 4 weeks premature

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change in proinflammatory miRNAs | Blood will be drawn before surgical incision, at the conclusion of the surgery (typically ~1 hour after incision), and at arrival to the PACU (typically 10-30 minutes after end of surgery)
  Blood samples will be analyzed for a composite measure of systemic inflammation caused by the anesthetic agent. MicroRNA (miRNA) expression will be compared between the time points for each patient and between arms.
  Total RNA will be extracted from whole blood using a commercially available kit. RNA will then be assayed for transcriptome analysis using microarray technology.
  Serum cytokines will be analyzed using Enzyme-Linked Immunosorbent Assay (ELISA) for Tumor Necrosis Factor alpha (TNF-α), Interleukin one beta (IL-1β),Monocyte Chemoattractant Protein one (MCP-1), Prostaglandin E2 (PGE2), Nuclear Factor kappa-light-chain-enhancer of activated B cells (NF-ĸB), transcription factor p65, and S100 calcium-binding protein B (S100B). miR-155, miR-146a, miR-146b, and miR-142-3p will be quantified using quantified polymerase chain reaction (qPCR).

SECONDARY OUTCOMES:
Change in systemic inflammation | Blood will be drawn before surgical incision, at the conclusion of the surgery (typically ~1 hour after incision), and at arrival to the PACU (typically 10-30 minutes after end of surgery)
  Inflammatory biomarkers in the serum will be compared between time points and between arms.